CLINICAL TRIAL: NCT05439772
Title: Examining the Effect of Ondansetron on Bowel Prep Success
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York - Downstate Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1650686-6
Record Dates: First submitted 2022-06-23; First posted 2022-06-30 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Abdominal Pain; Inflammatory Bowel Diseases; Eosinophilic Gastroenteritis; Diarrhea; Hematochezia; Weight Loss
Keywords: colonoscopy; bowel preparation; ondansetron
MeSH Terms: conditions — Abdominal Pain; Inflammatory Bowel Diseases; Eosinophilic enteropathy; Diarrhea; Gastrointestinal Hemorrhage; Weight Loss | interventions — Ondansetron

STUDY DESIGN:
Intervention Model Description: non-blinded randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Pediatric patients between the ages of 2-20 who have a clinical indication for colonoscopy, who will undergo standard colonoscopy preparation of polyethylene glycol and bisacodyl
- Ondansetron (Experimental): Pediatric patients between the ages of 2-20 who have a clinical indication for colonoscopy, who will undergo standard colonoscopy preparation of polyethylene glycol and bisacodyl with the addition of one dose of ondansetron prior to initiating bowel preparation.
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Ondansetron — Patient will take one dissolvable tablet of ondansetron prior to initiating PEG consumption.
  Other Names: Zofran
  Arms: Ondansetron

SUMMARY:
This is a pilot randomized-controlled trial assessing the utility of ondansetron for improving pediatric pre-colonoscopy bowel prep outcomes using the boston bowel preparation score, as well as assessing the impact on patient experience of bowel preparation.

DETAILED DESCRIPTION:
The study will compare two approaches to pre-colonoscopy cleanout, one with traditional laxatives only, and one with laxatives + anti-emetic therapy. The medication to be added will be Ondansetron (brand name: Zofran). Classically, the bowel prep entails drinking large amounts of water with an osmotic laxative and being only on a liquid diet the day prior to the procedure. Drinking this mixture of water with an osmotic laxative may cause nausea and discomfort in some patients that may prevent them from finishing the bowel prep. This will therefore affect the visualization of the colon during the procedure, as there will still be retained, hard stool. Having large amounts of stool in the colon during the procedure can make the colonoscopy more difficult, takes a longer time to complete, can make the study inconclusive, unable to properly diagnose, and difficult to take biopsies. This study assesses the impact of anti-emetic medication (ondansetron) on the bowel prep experience with the goal of improving participant tolerance and preparation success. This will eliminate concern for retained stool and less chance of cancelling a procedure due to improper bowel prep.

ELIGIBILITY:
Inclusion Criteria:

* Age >2, <20
* clinically indicated for a colonoscopy

Exclusion Criteria:

* known arrhythmia or long QT

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Boston Bowel Preparation Scale | 24 hours after dose
  validated scoring system of bowel preparation

SECONDARY OUTCOMES:
Symptoms associated with Bowel Prep | 24 hours after dose
  assess participant reports of pain, bloating, nausea, and vomiting associated with bowel preparation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wallach, MD, Principal Investigator — SUNY Downstate HSU
Locations (1):
- SUNY Downstate University Hospital of Brooklyn, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arostegui D, Armaly P, Castro Ochoa K, Lemus VV, Peshimam J, Sharma S, Schwarz S, Wallach T. Pilot Study of Ondansetron in Improvement of Pediatric Colonoscopy Preparation Outcomes at an Urban Academic Center. JPGN Rep. 2023 Sep 8;4(4):e366. doi: 10.1097/PG9.0000000000000366. eCollection 2023 Nov. PMID 38034452